CLINICAL TRIAL: NCT00297375
Title: A Comparison of the Efficacy and Safety of ULTRACET® (Tramadol HCl/Acetaminophen) Versus Placebo for the Acute Treatment of Migraine Headache Pain
Brief Title: A Study Comparing the Effectiveness and Safety of ULTRACET® (Tramadol HCl/Acetaminophen) Versus Placebo for the Treatment of Acute Pain From a Migraine Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002821
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Migraine; Head Pain; Headache
Keywords: treatment; Pain; acute; migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache; Pain

INTERVENTIONS:
Drug: tramadol HCl/acetaminophen

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of tramadol HCl/acetaminophen as a pain medication compared with placebo in the treatment of acute pain from a migraine headache. Although tramadol HCl/acetaminophen is approved to treat acute pain, it is not approved for the treatment of acute pain associated with migraine headache. The study hypothesis is that tramadol HCl/acetaminophen is safe and effective as a pain medication in the treatment of acute pain associated with a migraine headache.

DETAILED DESCRIPTION:
Although new drugs and procedures are available to treat acute migraine pain, inadequacies in treatment still exist. The ingredients in tramadol HCl/acetaminophen tablet and the way it works may be effective in the treatment of the pain of acute migraine headache. The combination of tramadol HCl/ acetaminophen works faster than tramadol alone and lasts longer than acetaminophen alone. This is a multicenter, single-dose, outpatient, randomized (study with two groups one in treatment and one control group), double-blind (neither patient nor investigator knows which patient is receiving study drug or control treatment), placebo-controlled, parallel-group (each group receives only one type of treatment) study of adult patients who experience at least moderate pain from migraine headaches. After being randomly assigned to a group patients will leave the study center with one dose (2 tablets) of study medication, either active treatment or placebo. The next time the patient has a migraine headache of at least moderate pain, the patient will take the study medication and start to answer questions about their headache pain and pain relief in a study diary. Patients should return to the study center within 72 hours of taking this dose. The study hypothesis is that tramadol HCl/acetaminophen is safe and effective as a pain medication in the treatment of acute pain associated with a migraine headache.

2 tramadol HCl (37.5 milligrams)/acetaminophen (325 milligrams) combination tablets or 2 matching placebo (inactive substance) tablets for tramadol HCl/acetaminophen taken one time orally

ELIGIBILITY:
Inclusion Criteria:

* Patient with a history of diagnosis of migraine with or without a warning sign (aura), that meets the criteria for a migraine, for at least 1 year
* History of migraine pain at least moderate in intensity
* Incidence of 1 to 6 headaches per month in the past year
* If female, using acceptable method of birth control

Exclusion Criteria:

* Patients with routine headaches that could be confused with migraines
* No more than 13 headache days per month in the past 6 months
* Onset of migraines after age 50
* Patients with migraines involving the eyes, chronic migraine or cluster headaches
* Patients using one or more of the following medications before study entry: more than 1 type of migraine prevention medicine in the past 6 weeks, tramadol within 30 days, vitamins/herbal remedies or non-drug-related remedies for migraine for < 30 days, St. John's Wort within 30 days, investigational drug in past 30 days or any other disallowed medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2003-04; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change in baseline headache pain severity at 2 hours post-dose from severe or moderate to mild or none, without using any nausea medication or other pain medication

SECONDARY OUTCOMES:
Pain free at 2, 6 and 24 hrs post-dose; difference in pain intensity and response to therapy over the first 6 hrs post-dose; reduction in occurrence and severity of symptoms; change in functional disability; subject overall rating of change.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Silberstein SD, Freitag FG, Rozen TD, Kudrow DB, Hewitt DJ, Jordan DM, Fisher AC, Rosenthal NR; CAPSS-223 Investigators. Tramadol/acetaminophen for the treatment of acute migraine pain: findings of a randomized, placebo-controlled trial. Headache. 2005 Nov-Dec;45(10):1317-27. doi: 10.1111/j.1526-4610.2005.00264.x. PMID 16324164
- See also: A Comparison of the Efficacy and Safety of ULTRACET® (Tramadol HCl/Acetaminophen) versus Placebo for the Acute Treatment of Migraine Headache Pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=492&filename=CR002821_CSR.pdf